CLINICAL TRIAL: NCT01266733
Title: Improvement of the Health-related Quality of Life of Patients With Fibromyalgia Using Multidisciplinary Treatment
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hospital Galdakao-Usansolo (Other Government)
Responsible Party: Principal Investigator, Josune Martin Corral, PhD, Hospital Galdakao-Usansolo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2006111057
Record Dates: First submitted 2010-12-23; First posted 2010-12-24 (Estimated); Last update posted 2015-06-18 (Estimated); Status verified 2010-12

CONDITIONS: Fibromyalgia
Keywords: fibromyalgia, non pharmacological intervention
MeSH Terms: conditions — Fibromyalgia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Interdisciplinary treatment (Experimental)
  Interventions: Behavioral: Interdisciplinary treatment; Behavioral: Interdisciplinary treatment of fibromyalgia
- Usual treatment (No Intervention)

INTERVENTIONS:
Behavioral: Interdisciplinary treatment — The Experimental Group received 6 weeks of interdisciplinary treatment of fibromyalgia combining coordinated psychological, medical, educational, and physiotherapeutic interventions delivered by a team that included a physician, a psychologist, and a physiotherapist.Patients in the EG were divided into groups of 12 individuals. Each attended biweekly group sessions of 1 hour and 45 minutes, for a total of 12 sessions. One session included 1 hour with the psychologist and 45 minutes of educational activities with the physician and psychologist, while the other session included 1 hour with the psychologist and 45 minutes with the physiotherapist.
  Other Names: Interdisciplinary treatment of fibromyalgia
  Arms: Interdisciplinary treatment
Behavioral: Interdisciplinary treatment of fibromyalgia — The Control Group received the usual standard of care, which included pharmacologic treatment with a tricyclic antidepressant (amitriptyline, maximum dose of 75 mg/24h), an analgesic (paracetamol, maximum dose of 4 grams/24h), and a non-opioid central analgesic (tramadol, maximum dose of 400 mg/24h). The Experimental Group (EG) received 6 weeks of interdisciplinary treatment combining coordinated PSYchological, Medical, Educational, and PHYsiotherapeutic interventions (PSYMEPHY) delivered by a team that included a physician, a psychologist, and a physiotherapist. Patients in the EG were divided into groups of 12 individuals. Each attended biweekly group sessions of 1 hour and 45 minutes, for a total of 12 sessions.
  Arms: Interdisciplinary treatment

SUMMARY:
The purpose of this study is to assess improvement in health related quality of life of fibromyalgia patients following 6 weeks of interdisciplinary treatment compared to the usual treatment.

DETAILED DESCRIPTION:
Fibromyalgia (FM) is the most common cause of diffuse pain in the bones and joints, with a prevalence in general adult populations estimated at between 0.7% and 3.3%. In Spain, the prevalence of FM is 2-3%; it affects mainly women, with new diagnoses peaking between the ages of 40 and 49 years. In certain populations, however, the prevalence may be much higher, as in 15% of patients referred from internal medicine units or 12% of patients referred to rheumatology specialists in Spain.

Fibromyalgia produces various degrees of disability and pain. It also has a clear impact on health-related quality of life (HRQoL). Burckhardt et al. observed lower HRQoL among patients with fibromyalgia than among healthy subjects. Indeed, the HRQoL for those with FM was similar to that of patients with insulin-dependent diabetes mellitus or chronic obstructive pulmonary disease. Among patients with non-cancer chronic pain referred to the pain management unit at our institution, those with bone and joint pain and with FM had the worst progress 6 months after diagnosis as measured by HRQoL.

The characteristics of FM, such as its complex and unknown etiology, wide range of symptoms and signs, and multiple comorbidities make identifying effective therapies particularly difficult. As a result, no consensus yet exists regarding the best therapeutic approaches, and treatment of FM presents a challenge for clinicians. Clinical research suggests that pharmacologic treatment alone is not the best approach for FM, and that an integrated biopsychosocial approach that includes non-pharmacologic therapies along with pharmacologic therapies improves outcomes in these patients.

In our hospital, between 5% and 10% of patients newly diagnosed with FM are referred to the pain management unit. We established a clinical trial in this population to assess improvement in HRQoL following 6 months of interdisciplinary treatment compared to the usual treatment, as well as to identify predictors for improvement in HRQoL.

ELIGIBILITY:
Inclusion Criteria:

* a patient must have been diagnosed with FM according to diagnostic criteria of the American College of Rheumatology
* being 18 years or older and
* having had continuous chronic pain for at least 6 months.

Exclusion Criteria:

* Patients were excluded if they did not agree to participate in the study,
* were suffering from a severe psychiatric or organic disorder, or
* were involved in employment-related legal proceedings related to their FM. Participants in the trial were required to sign an informed consent form.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 153 (Actual)
Dates: Start 2007-02; Primary Completion 2009-12 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Health-related quality of life among patients with fibromyalgia (FIQ: Fibromyalgia Impact Questionnaire) | 6 months
  Fibromyalgia patients completed the FIQ at baseline and again 6 months after the interdisciplinary intervention.

SECONDARY OUTCOMES:
Anxiety and depressive symptoms (HADS: The Hospital Anxiety and Depression Scale) | 6 months
  Patients with fibromyalgia completed the HADS at baseline and again 6 months after the intervention

CONTACTS AND LOCATIONS:
Overall Officials: Fernando Torre, Doctor, Principal Investigator — Hospital Galdakao-Usansolo (Bizkaia) Spain
Locations (1):
- Hospital Galdakao-Usansolo, Galdakao, Bizkaia, Spain

REFERENCES:
- [Derived] Martin J, Torre F, Padierna A, Aguirre U, Gonzalez N, Matellanes B, Quintana JM. Impact of interdisciplinary treatment on physical and psychosocial parameters in patients with fibromyalgia: results of a randomised trial. Int J Clin Pract. 2014 May;68(5):618-27. doi: 10.1111/ijcp.12365. Epub 2014 Feb 20. PMID 24868587